CLINICAL TRIAL: NCT03876886
Title: Randomized Phase Ⅲ Trial Comparing Dose-dense Epirubicin and Cyclophosphamide Followed by Paclitaxel With Paclitaxel Plus Carboplatin as Adjuvant Therapy for Triple-negative Breast Cancer With Homologous Recombination Repair Deficiency
Brief Title: The Trial Comparing Dose-dense AC-T With TP as Adjuvant Therapy for TNBC With Homologous Recombination Repair Deficiency
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Binghe Xu, Professor of Medical Oncology, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BXu-1839
Record Dates: First submitted 2019-03-14; First posted 2019-03-15 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Triple Negative Breast Cancer
Keywords: homologous recombination deficiency;adjuvant chemotherapy;anthracycline;taxanes;platinum
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Epirubicin; Cyclophosphamide; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AC-T(dose-dense) (Active Comparator): A: epirubicin, pharmorubicin (EPI) C: cyclophosphamide (CTX） T: paclitaxel (PTX）
  Interventions: Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Paclitaxel
- TP(dose-dense) (Experimental): T: paclitaxel (PTX） P: carboplatin (CBP)
  Interventions: Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Epirubicin — Epirubicin 90mg/m2 iv d1 or divide into two days
  Arms: AC-T(dose-dense)
Drug: Cyclophosphamide — cyclophosphamide600mg/m2 iv d1,q14d*4cycles;with G-CSF support: 3ug/kg ih
  Arms: AC-T(dose-dense)
Drug: Paclitaxel — paclitaxel 175mg/m2 iv d1, q14d*4cycles
  Arms: AC-T(dose-dense)
Drug: Carboplatin — carboplatin AUC=3 iv d2, q14d*8cycles;with G-CSF support: 3ug/kg ih
  Arms: TP(dose-dense)
Drug: Paclitaxel — paclitaxel 175mg/m2 iv d1, q14d*8cycles
  Arms: TP(dose-dense)

SUMMARY:
The purpose of this trial is to compare the 3-year disease-free survival of dose-dense epirubicin and cyclophosphamide followed by paclitaxel with paclitaxel plus carboplatin as adjuvant therapy for triple-negative breast cancer with homologous recombination repair deficiency.

The other purpose of this trial is to observe the patient's tolerance.

DETAILED DESCRIPTION:
Triple-negative breast cancer (TNBC) lack the expression of oestrogen receptor (ER), progesterone receptor(PR) and human epidermal growth factor receptor 2 (HER2) , and characterizes an aggressive behavior with higher risk of recurrence and death compared to other breast cancer subtypes. Little therapeutic progress has been made in adjuvant therapy in TNBC during the past decades and the standard of care is still missing.

Pre-clinical and clinical data suggest that platinum-based regimens represent an emerging therapeutic option for selected patients with homologous recombination repair deficiency (HRD). The HR system is critical in regulating and maintaining genome stability, and is one of the most commonly altered systems in TNBCs, up to 15-20% TNBC patients carry germline BRCA1/2 mutations. Other HR genes included PALB2, RAD51 etc. Tumors that harbor HRD possess an increased burden of genomic aberrations and lesions, and have been shown to have increased sensitivity to DNA crosslinking agents such as platinum salts. Platinum-based regimens have been encouraging in TNBC patients with HRD, given increases in both pathologic complete response (pCR) rates in neoadjuvant trials and objective response rates(ORR) in metastatic diseases. Further information are needed on how platinum-containing therapies affect long-term outcomes in the adjuvant setting.

In this trial, the investigators intend to compare the 3-year disease-free survival (DFS) of dose-dense epirubicin and cyclophosphamide followed by paclitaxel with paclitaxel plus carboplatin as adjuvant therapy in high-risk node-negative or node-positive TNBC patients with HRD. The other purpose of this trial is to observe the participants' tolerance.

ELIGIBILITY:
Inclusion Criteria:

1. 18-60 years
2. Histologically confirmed adenocarcinoma of the breast, complete tumor removal by either modified radical mastectomy or local excision plus axillary lymph node dissection (i.e., breast conservation therapy) or sentinel node biopsy. (Tumor-free margins at least 1 mm for both invasive and noninvasive carcinoma except for lobular carcinoma in situ (less than 1 mm allowed);
3. Histologically confirmed ER(-) PR(-) and HER-2(IHC(immunohistochemistry) 0-1+ or FISH (fluorescence in situ hybridization) negative)
4. Next-generation sequencing confirmed homologous recombination repair deficiency
5. Meet one of the following criteria:

(1) Positive axillary lymph nodes; (2) Negative axillary lymph nodes with at least one of the following risk factors: age<= 35 years; grade III; infiltrative tumor size > 2cm; intravascular tumor embolus; Ki-67>=50%.

6. Eastern Cooperative Oncology Group (ECOG) Performance Score 0-1 7. Adequate bone marrow reserve with ANC > 1500, HGB > 9g/dL and platelets > 100,000.

8. Adequate renal function with serum creatinine < 2.0. 9. Adequate hepatic reserve with serum bilirubin < 2.0, AST/ALT < 2X the upper limit of normal, and alkaline phosphatase < 5X the upper limit of normal. Serum bilirubin > 2.0 is acceptable in the setting of known Gilbert's syndrome.

10. Not pregnant, and on appropriate birth control if of child-bearing potential.

11. Written informed consent according to the local ethics committee requirements.

Exclusion Criteria:

1. Prior systemic treatment of breast cancer, including chemotherapy;
2. Metastatic breast cancer;
3. Patients with medical conditions that indicate intolerant to adjuvant therapy and related treatment, including uncontrolled pulmonary disease, diabetes mellitus, severe infection, active peptic ulcer, coagulation disorder, connective tissue disease or myelo-suppressive disease;
4. Has active hepatitis B or hepatitis C with abnormal liver function tests (LFTs) or is known to be HIV positive;
5. Contraindication for using dexamethasone;
6. History of congestive heart failure, uncontrolled or symptomatic angina pectoris, arrhythmia or myocardial infarction; poorly controlled hypertension (systolic BP>180 mmHg or diastolic BP>100 mmHg);
7. Pregnant or breast feeding.
8. Hepatic, renal, or bone marrow dysfunction as detailed above.
9. Known severe hypersensitivity to any drugs in this study;
10. Treatment with any investigational drugs within 30 days before the beginning of study treatment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-02-22 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
3-year disease-free survival | Three years
  The participants will be followed by the telephone for the duration, an expected average of 3 years.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Three years
  Incidence of neutropenic fever; Incidence of grade 3-4 side effects; Toxicity assessed by NCI CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center, Cancer Hospital/Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China